CLINICAL TRIAL: NCT07000461
Title: Can Transcranial Doppler Predict Postoperative Cognitive Dysfunction After Cardiopulmonary Bypass
Brief Title: Transcranial Doppler as a Predictor of Postoperative Cognitive Dysfunction Following Cardiopulmonary Bypass
Status: Recruiting | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025/102
Record Dates: First submitted 2025-04-16; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Cognitive Dysfunction; Delirium, Postoperative
Keywords: transcranial doppler; delirium; POCD; cerebral perfusion; CABG
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Pulsatile perfusion: Pulsatile group in pump blood flow
  Interventions: Procedure: Group Non-pulsatile perfusion

INTERVENTIONS:
Procedure: Group Non-pulsatile perfusion — Non-pulsatile group in pump blood flow

SUMMARY:
Neurological dysfunction either transient or permanent is a major cause of morbidity and mortality after cardiopulmonary bypass, and cognitive dysfunction is more frequent in cardiac surgery than in non-cardiac procedures. Variations in cerebral blood flow and oxygen extraction are considered key contributing factors. Although pulsatile flow during bypass has shown benefits for renal function and recovery, its effects on postoperative neurological dysfunction and delirium remain unclear due to limited research. This study aims to evaluate the impact of pulsatile versus non-pulsatile cardiopulmonary bypass flow on POCD in adult CABG patients by measuring middle cerebral artery (MCA) flow using transcranial Doppler.

DETAILED DESCRIPTION:
Patient Selection:

Our study is a single-center, prospective, observational study. The study will include 65 patients scheduled for elective coronary artery bypass grafting (CABG) surgery between 01.04.2025 and 31.03.2026 at the Health Sciences University, Bakırköy Dr. Sadi Konuk Training and Research Hospital. Patients aged 18-70, and those scheduled for isolated elective coronary artery bypass grafting, will be included. Patients with carotid stenosis greater than 50%, a history of cerebrovascular events, those who do not provide consent, those with temporal window failure, ejection fraction (EF) below 40%, a preoperative Mini-Mental State Examination (MMSE) score under 23, those requiring mechanical ventilation for more than 24 hours, or those requiring reintubation will be excluded from the study.

Preoperative Preparation:

Patients eligible for the study will be informed about the study, and a voluntary consent form will be obtained. The demographic characteristics of the patients (age, gender, comorbidities, ASA score, BMI, ejection fraction, kidney function tests, EUROSCORE 2 score) will be recorded. All patients will undergo the Mini-Mental State Examination (MMSE) 24 hours before the operation. All patients will undergo standard cardiovascular surgical monitoring (electrocardiography (ECG), non-invasive blood pressure monitoring, peripheral oxygen saturation (SpO2), bilateral regional cerebral oxygen saturation (rSO2) measured by near-infrared spectroscopy (NIRS), and processed EEG monitoring). At the beginning of anesthesia, two 18-20 G granule peripheral venous access lines will be established. The decision regarding whether to use pulsatile or non-pulsatile pump flow will be made by the surgical team. The preoperative baseline (T1) middle cerebral artery (MCA) flow value will be measured using transcranial Doppler with a low-frequency (2-3.5 MHz) sector/cardiac probe. The trans-temporal window, one of the acoustic windows of the skull, will be identified anatomically by locating the hyperechoic image of the sphenoid and temporal bone petrous part between the upper zygomatic arch, external auditory canal, and orbit. In the color Doppler mode of ultrasound, MCA flow will be observed at a depth of 3-7 cm with the probe approaching, and pulse wave (PW) Doppler will be applied. Peak systolic and end-diastolic measurements will be recorded as the average of the three values shown on the screen and documented. Invasive arterial monitoring will be routinely performed.

Perioperative Process:

During anesthesia induction, patients will receive 0.1-0.2 mg/kg of midazolam, 5-8 µg/kg of fentanyl, and 0.6 mg/kg of rocuronium. Anesthesia depth will be maintained with sevoflurane inhalation, dexmedetomidine, and remifentanil infusion, with a Patient State Index (PSI) general anesthesia level maintained between 25-50. After anesthesia induction (T2), after cross-clamping at the 10th minute (T3), 20th minute (T4), 30th minute (T5), after the cross-clamp is removed (T6), and at the end of surgery (T7), transcranial Doppler measurements, mean arterial pressure (MAP), and cerebral oxygen saturation (rSO2) values will be recorded. Arterial blood gas analyses will be recorded at T2, T3, T6, and T7.

Postoperative Process :

The patient will be admitted to the Postoperative Cardiovascular Surgery Intensive Care Unit. At 24 hours postoperatively, delirium will be assessed using the CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) in the intensive care unit. For patients with prolonged ICU stays, delirium assessments using CAM-ICU will continue. On the 2nd-4th days, delirium evaluation will be conducted in the morning and evening using the 3DCAM test in the service setting. At 24 hours, ventilator time, fluid balance, urine output, inotropic/vasopressor requirements, presence of new arrhythmias, amount of blood products used postoperatively, kidney function tests (AKI), and other recorded data will be evaluated. A repeat Mini-Mental State Examination (MMSE) will be performed on the 5th day of the hospital stay. Cerebrovascular events during the hospital stay will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70
* Patients scheduled for isolated elective cardiopulmonary bypass surgery

Exclusion Criteria:

* Patients with carotid stenosis ≥50%
* Emergency patients or those with a history of reoperation
* Patients with a history of cerebrovascular events
* Patients who do not provide consent
* Patients with temporal window failure
* Patients with an ejection fraction (EF) <40%
* Patients with a Mini-Mental State Examination (MMSE) score <23
* Patients who require mechanical ventilation for more than 24 hours or those who are reintubated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for isolated elective cardiopulmonary bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative Cerebral Perfusion | pre anesthesia induction
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.
Perioperative Cerebral Perfusion | post anesthesia induction
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.
Perioperative Cerebral Perfusion | 10th minute after aortic cross-clamp
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.
Perioperative Cerebral Perfusion | 20th minute after aortic cross-clamp
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.
Perioperative Cerebral Perfusion | 30th minute after aortic cross-clamp
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.
Perioperative Cerebral Perfusion | remove cross-clamp
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.
Perioperative Cerebral Perfusion | end of the surgery
  Perioperative transcranial doppler will be used to measure middle cerebral artery flow.

SECONDARY OUTCOMES:
Acute kidney injury | Postoperative 24th hour
  Postoperative 24th hour urea creatine value and urine output
Duration of mechanical ventilation | Postoperative 24th hour
  The duration of ventilator support withdrawal in the postoperative intensive care unit
Length of stay in intensive care | within 30 days after surgery
  The time the patient is transferred from intensive care to the ward
Length of hospital stay | within 60 days after surgery
  The time the patient is discharged home

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided